CLINICAL TRIAL: NCT02510365
Title: Safety and Efficacy of Functional Neural Regeneration Collagen Scaffold Transplantation in Complete (AISA) Acute Spinal Cord Injury Patients
Brief Title: Functional Neural Regeneration Collagen Scaffold Transplantation in Acute Spinal Cord Injury Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Affiliated Hospital of Logistics University of CAPF (Other); The First Affiliated Hospital of Soochow University (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); General Hospital of Ningxia Medical University (Other); Army Medical University, China (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAS-XDA-ACSCI/IGDB
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2015-07

CONDITIONS: Acute Spinal Cord Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional collagen scaffold (Experimental): Functional neural regeneration collagen scaffold transplantation.
  Interventions: Biological: Functional collagen scaffold

INTERVENTIONS:
Biological: Functional collagen scaffold — Patients will receive functional neural regeneration collagen scaffold and patients will undergo a comprehensive rehabilitation and psychological measures after surgery.

SUMMARY:
The study is designed to assess the safety and efficacy of functional neural regeneration collagen scaffold transplanted into acute spinal cord injury patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years old.
2. Completely spinal cord injury at the cervical and thoracic level (C4-T12).
3. Classification ASIA A, occurring within past 21 days.
4. Patients signed informed consent.
5. Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.

Exclusion Criteria:

1. A current diagnosis of any primary diseases affecting limb functions (e.g., trauma, infection, tumors, congenital malformations, peripheral muscular dystrophy, Huntington's disease, Parkinson's disease).
2. Serious complications (e.g., hydronephrosis due to renal insufficiency, severe bedsores (Ⅲ° above), lower extremity venous thrombosis, severe myositis ossificans).
3. History of life threatening allergic or immune-mediated reaction.
4. Clinically significant abnormalities in routine laboratory examinations (hematology, electrolytes, biochemistry, liver and kidney function tests, urinanalysis).
5. History of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
6. Severe arrhythmias (e.g., ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
7. Lactating and pregnant woman.
8. Alcohol drug abuse /dependence.
9. Participated in any other clinical trials within 3 months before the enrollment.
10. A drug or treatment known to cause effect on the central nervous system during the past four weeks.
11. A drug or treatment known to cause major organ system toxicity during the past four weeks.
12. Poor compliance, difficult to complete the study.
13. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation Number of patients with adverse events | 6 months
  Number of patients with adverse events is as a measure of safety and tolerability after collagen scaffold transplantation.

SECONDARY OUTCOMES:
Improvements in ASIA Impairment Scale | 12 months
  American Spinal Injury Assessment Scale of A, B, C, D or E will be assessed before and after transplantation.
Improvements in Electrophysiological monitoring | 12 months
  Somatosensory Evoked Potentials (SSEP) monitoring will be assessed before and after transplantation.
Improvements in Electrophysiological monitoring | 12 months
  Motor Evoked Potentials (MEP) monitoring will be assessed before and after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences; Sai Zhang, M.D, Study Chair — Affiliated Hospital of Logistics Universtiy of CAPF; Huilin Yang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University; Shuxun Hou, Study Chair — First Hospitals affiliated to the China PLA General Hospital; Hechun Xia, Study Chair — General Hospital of Ningxia Medical University; Tongwei Chu, Study Chair — Army Medical University, China
Locations (5):
- China (5):
  - First Hospitals affiliated to the China PLA General Hospital, Beijing
  - Xinqiao Hospital of Army Medical University, Chongqing
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Affiliated Hospital of Logistics Universtiy of CAPF, Tianjin
  - General Hospital of Ningxia Medical University, Yinchuan

REFERENCES:
- [Derived] Chen W, Zhang Y, Yang S, Sun J, Qiu H, Hu X, Niu X, Xiao Z, Zhao Y, Zhou Y, Dai J, Chu T. NeuroRegen Scaffolds Combined with Autologous Bone Marrow Mononuclear Cells for the Repair of Acute Complete Spinal Cord Injury: A 3-Year Clinical Study. Cell Transplant. 2020 Jan-Dec;29:963689720950637. doi: 10.1177/0963689720950637. PMID 32862715
- [Derived] Xiao Z, Tang F, Zhao Y, Han G, Yin N, Li X, Chen B, Han S, Jiang X, Yun C, Zhao C, Cheng S, Zhang S, Dai J. Significant Improvement of Acute Complete Spinal Cord Injury Patients Diagnosed by a Combined Criteria Implanted with NeuroRegen Scaffolds and Mesenchymal Stem Cells. Cell Transplant. 2018 Jun;27(6):907-915. doi: 10.1177/0963689718766279. Epub 2018 Jun 5. PMID 29871514